CLINICAL TRIAL: NCT00071331
Title: Protocol 156-03-236: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Long Term Efficacy and Safety of Oral Tolvaptan Tablets in Subjects Hospitalized With Worsening Congestive Heart Failure
Brief Title: EVEREST: Efficacy of Vasopressin Antagonism in hEart failuRE: Outcome Study With Tolvaptan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-03-236
Record Dates: First submitted 2003-10-20; First posted 2003-10-21 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Congestive Heart Failure
Keywords: chronic heart failure; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan

SUMMARY:
The purpose of this study is to compare the effectiveness of tolvaptan or placebo in adults with worsening congestive heart failure (CHF).

DETAILED DESCRIPTION:
Study Design: Multicenter, randomized, double-blind, placebo-controlled

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Current hospitalization for chronic congestive heart failure with admission up to 48 hours prior to randomization. Chronic heart failure is defined as requiring treatment for a minimum of 30 days prior to hospitalization.

The subject must have signs of extracellular volume expansion, defined as two or more of the following: a) jugular venous distention; b) pitting edema (>1+); or c) dyspnea.

* NYHA Class III or IV at the time of hospitalization.
* Left Ventricular Ejection Fraction < = 40% within one year.

Exclusion Criteria

* Women who will not adhere to the reproductive precautions as outlined in the Informed Consent form.
* Positive urine pregnancy test.
* Inability to provide written informed consent.
* Cardiac surgery within 60 days of potential study enrollment, excluding percutaneous coronary interventions.
* Planned revascularization procedures, electrophysiologic (EP) device implantation, cardiac mechanical support implantation, cardiac transplantation, or other cardiac surgery within 30 days following study enrollment.
* Subjects who are on cardiac mechanical support.
* History of bi-ventricular pacer placement within the last 60 days.
* Co-morbid condition with an expected survival less than six months.
* Subjects with acute ST segment elevation myocardial infarction at the time of hospitalization.
* History of sustained ventricular tachycardia or ventricular fibrillation within 30 days, unless in the presence of an automatic implantable cardioverter defibrillator.
* History of a cerebrovascular accident within the last 30 days.
* Hemodynamically significant uncorrected primary cardiac valvular disease.
* Hypertrophic cardiomyopathy (obstructive or non-obstructive).
* CHF due to uncorrected thyroid disease, active myocarditis or known amyloid cardiomyopathy.
* Subjects with progressive or episodic neurological disease such as multiple sclerosis or history of multiple strokes.
* History of primary significant liver disease or acute hepatic failure, as defined by the investigator.
* History of poorly controlled diabetes mellitus.
* Morbid obesity, defined as > 159 kg (or 350 lbs) or BMI > 40.
* Supine systolic arterial blood pressure < 90 mmHg.
* Serum creatinine > 3.5 mg/dL or > 309.4 mmol/L.
* Serum potassium > 5.5 mEq/L or > 5.5 mmol/L.
* Hemoglobin < 9 g/dL or < 90 g/L.
* History of hypersensitivity and/or idiosyncratic reaction to benzazepine derivatives (such as benazapril).
* History of drug or medication abuse within the past year, or current alcohol abuse.
* Inability to take oral medications.
* Participation in another clinical drug or device trial within the past 30 days.
* Previous participation in this or any other tolvaptan clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600
Dates: Start 2003-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (377):
- United States (160):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Heart Center, Huntsville, Alabama
  - The Heart Group, Mobile, Alabama
  - Phoenix Memorial Hospital, Gilbert, Arizona
  - Arizona Heart Institute, Phoenix, Arizona
  - Saguaro Clinical Research, Tucson, Arizona
  - Central Arkansas Veterans Healthcare Systems, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Central Cardiology Medical Center, Bakersfield, California
  - Cardiology Associates, Larkspur, California
  - Loma Linda University Medical Center, Loma Linda, California
  - LAC/USC Medical Center, Los Angeles, California
  - VA Medical Center- W. Los Angeles, Los Angeles, California
  - Mission Internal Medical Group, Mission Viejo, California
  - ARI Clinical Trials, Redondo Beach, California
  - San Diego Cardiac Center, San Diego, California
  - Pacific Heart Institute, Santa Monica, California
  - Cardiovascular Consultants Medical Group, Inc., Walnut Creek, California
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Heart and Vascular Clinic of North Colorado, Fort Collins, Colorado
  - Bakus Resesarch, Norwich, Connecticut
  - Christiana Care Health System, Newark, Delaware
  - VA Medical Center, Washington D.C., District of Columbia
  - Florida Cardiovascular Research, Atlantis, Florida
  - Cardiology Associates of Fort Lauderdale, Fort Lauderdale, Florida
  - Jacksonville Heart Center, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Heart Center, Jacksonville Beach, Florida
  - Melbourne Internal Medicine Assoc., Melbourne, Florida
  - University of Miami/ Jackson Memorial Hospital, Miami, Florida
  - Miami Research and Education Foundation, Miami, Florida
  - Ocala Resarch Institute, Ocala, Florida
  - Cardiology Research Associates, Ormond Beach, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - The Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Cardiac Disease Specialists PC, Atlanta, Georgia
  - Atlanta Heart and Vascular Research Group, Atlanta, Georgia
  - Georgia Heart Specialists, Covington, Georgia
  - Idaho Cardiology Associates, Boise, Idaho
  - Idaho Cardiology Associates, Meridian, Idaho
  - North Shore Cardiologists, Bannockburn, Illinois
  - Northwestern University, Chicago, Illinois
  - Midwest Heart Research Found., Lombard, Illinois
  - Illinois Heart & Lung Associates, Normal, Illinois
  - Heart Care Midwest, Peoria, Illinois
  - The Care Group, Indianapolis, Indiana
  - Mid America Cardiology, Kansas City, Kansas
  - Cardiovascular Associates, Louisville, Kentucky
  - Louisville Cardiology Medical Group, Louisville, Kentucky
  - The Louisiana Heart Center, Chalmette, Louisiana
  - Northshore Medical Research, Covington, Louisiana
  - Leonard J Chabert Medical Center, Houma, Louisiana
  - Lousiana State University Health Sciences Center, Shreveport, Louisiana
  - Cardiac Centers of LA, LLC, Shreveport, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Northeast Cardiology Associates, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - MidAtlantic Cardiovascular Associates, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Bel Air, Maryland
  - Shore Health System, Easton, Maryland
  - MidAtlantic Cardiovascular Associates, Towson, Maryland
  - Heart Associates, P.A., Towson, Maryland
  - MidAtlantic Cardiovascular Associates, Westminster, Maryland
  - Primary Care Cardiology Research, Ayer, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Medical Center, Boston, Massachusetts
  - John Dingell VA Medical Center, Detroit, Michigan
  - Nisus Research, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Beaumont Hospital, Troy, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Division of Cardiology, Rochester, Minnesota
  - Park Nicollet Heart Center, Saint Louis Park, Minnesota
  - Regions Hospital Cardiology Research, Saint Paul, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - VA Medical Center- Kansas City, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Heart Consultants, Omaha, Nebraska
  - New England Heart Institute, Manchester, New Hampshire
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Garden State Cardiology, Paramus, New Jersey
  - Albany Associates in Cardiology, Albany, New York
  - Cardiology Associates, P.C., Johnson City, New York
  - North Shore University Hospital, Manhasset, New York
  - St. Vincents Hospital and Medical Center, New York, New York
  - St. Lukes-Roosevelt Hospital Centers, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - SUNY, Syracuse, New York
  - South Bay Cardiovascular Associates, West Islip, New York
  - Buffalo Cardiology and Pulmonary Associates, Williamsville, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Alamance Regional Medical Center, Burlington, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke Cardiology Research, Durham, North Carolina
  - Pitt County Memorial Hospital, The Heart Center, Greenville, North Carolina
  - Hendersonville Cardiology, Hendersonville, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Clinical Research Limited, Canton, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Midwest Cardiology Research Foundation, Columbus, Ohio
  - The Dayton Heart Center, Dayton, Ohio
  - Cleveland Cardiovascular Research, Fairview Park, Ohio
  - North Ohio Research Limited, Lorain, Ohio
  - North Ohio Research Limited, Sandusky, Ohio
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Integris Heart Research Center, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, LTD, Sayre, Pennsylvania
  - Buxmont Cardiology Associates, PC, Sellersville, Pennsylvania
  - Cardiology Associates of West Reading, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph H. Johnson VAMC, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - The Chattanooga Heart Institute, Chattanooga, Tennessee
  - Cardiovascular Associates, Kingsport, Tennessee
  - Baptist Clinical Research Center, Memphis, Tennessee
  - Stern Cardiovascular Center, Memphis, Tennessee
  - Vanderbilt Clinical Trials Center, Nashville, Tennessee
  - The Cardiology Group, Tullahoma, Tennessee
  - Austin Cardiovascular Associates, Austin, Texas
  - Southeast Texas Cardiology Associates, Beaumont, Texas
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Cardiology Associates Covenant Medical Group, Lubbock, Texas
  - McAllen Heart Clinic, McAllen, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Wilford Hall Medical Center,, San Antonio, Texas
  - Scott & White Clinic Division of Cardiology, Temple, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - The Cardiovascular Group PC, Fairfax, Virginia
  - Inova Institute of Research, Falls Church, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - Cardiovascular Associates of Virginia, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Empire Health Services, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - CAMC Clinical Trials, Charleston, West Virginia
  - Wisconsin Center For Clinical Research, Elkhorn, Wisconsin
- Argentina (20):
  - Clinica Constituyentes de Moron, Buenos Aires
  - Clinica Modelo de Moron, Buenos Aires
  - Fundacion Favaloro, Buenos Aires
  - Hospital Argerich, Buenos Aires
  - Hospital Churruca, Buenos Aires
  - Hospital Eva Peron, Buenos Aires
  - Hospital Nacional Dr. Alejandro Posadas, Buenos Aires
  - Hospital de Clinicas, Capital Federal
  - Hospital Fernandez, Capital Federal
  - Hospital Italiano de Buenos Aires, Capital Federal
  - Hospital Privado Antartida, Capital Federal
  - Hospital Ramos Mejia, Capital Federal
  - Policlinica Bancaria, Capital Federal
  - Sanatorio Municipal "Julio A. Mendez", Capital Federal
  - Instituto de Cardiologia J. F. Cabral, Corrientes
  - Hospital Allende, Córdoba
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Militar de Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Central de San Isidro, San Isidro
- Belgium (4):
  - AZ Middelheim, Antwerp
  - AZ Imelda Ziekenhuis, Bonheiden
  - Clinique St Elisabeth Place Louise, Namur
  - Cliniques UCL Mont-Godinne, Yvoir
- Brazil (19):
  - Hospital Santa Isabel da Santa Casa de Misericordia da Bahia, Salvador, Estado de Bahia
  - Fundacao Bahiana de Cardiologia- Hospital Universitario Professor Edgard Santos, Salvador, Estado de Bahia
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Governador Israel Pinheiro, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Evangelico de Curitiba, Curitiba, Paraná
  - Hospital Nossa Senhora das Gracas, Curitiba, Paraná
  - Santa Casa de Misericordia do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceica, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro, Campinas, São Paulo
  - Hospital de Base da Faculdade de Medicina de Sao Jose do Rio Preto, Sao Jose de Rio Preto, São Paulo
  - IMC- Instituto de Molestias Cardiovasculares, São José do Rio Preto, São Paulo
  - Instituto do Coracao do Hospital das Clinicas- Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital Universitario Onofre Lopes, Natal
  - Hospital das Clínicas de Porto Alegre, Porto Alegre
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro
- Canada (20):
  - Peter Loougheed Center, Calgary, Alberta
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Center, St. John's, Newfoundland and Labrador
  - Brampton Research Associates, Brampton, Ontario
  - Greater Niagara General Hospital, Niagara Falls, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Cardiology Research Associates, Scarborough Village, Ontario
  - The Scarborough Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto Western Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Sherbrooke, Fleurimond, Quebec
  - CHRDL, Joliette, Quebec
  - Invascor Clinical Research, Longueuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Hotel-Dieu de Saint-Jerome, Saint-Jérôme, Quebec
- Czechia (13):
  - I. interni kardio-angiologicka klinika LF MU, Brno
  - Interni oddeleni, Jablonec nad Nisou
  - Interni oddeleni, Náchod
  - Interni klinika, Oddeleni Interna I, Kardiologie, Pardubice
  - Interni oddeleni, Písek
  - I.Interni klinika, Plzen-Lochotin
  - I.Interni oddeleni, Prague
  - II.Interni klinika, Prague
  - Kardiologicka klinika, Prague
  - Kardiologicke oddeleni, Prague
  - Klinika kardiologie, Prague
  - Interni oddeleni, Ústí nad Labem
  - Interni klinika IPVZ, Zlín
- France (12):
  - Centre Hospitalier Regional d'Arras-Service de Cardiologie, Arras
  - Hopital General Henri Duffaut, Avignon
  - Centre Hospitalier Jeanne d'Arc, Bar-le-Duc
  - Hopital Louis Pradel, Bron
  - Cabinet de Cardiologie et d'Explorations, Essey-lès-Nancy
  - Centre Hospitalier, Langres
  - CHU Montpellier, Montpellier
  - Centre Hospitalo-Universitaire de Nantes-Service de Cardiologie, Nantes
  - Hopital Pasteur, Nice
  - Centre Cardiologique du Nord, Saint-Denis
  - Groupe Hospitalier Rangueil-Larrey CHU, Toulouse
  - Centre Hospitalier Universitaire de Nancy-Brabois, Vandœuvre-lès-Nancy
- Germany (21):
  - Klinikum Augsburg, Augsburg
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Herz- und Gefabklinik Bad Neustadt, Bad Neustadt-Saale
  - Vivantes Klinikum Neukoln, Berlin
  - Klinikum der Universitat zu Koln, Cologne
  - Akademisches Lehrkrankenhaus d. HGS Essen, Essen
  - Universitatsklinik Essen, Essen
  - Georg-August-Universitat Gottingen, Göttingen
  - Universitatsklinikum der, Greifswald
  - Klinikum der Medizinischen Fakultat, Halle
  - Universitatsklinikum Eppendorf, Hamburg
  - Medizinische Universitätsklinik, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum des Saarland, Homburg/Saar
  - Friedrich Schiller Universitat Jena, Jena
  - University Leipzig, Leipzig
  - Universitatsklinikum Munster, Münster
  - Herz- und Diabetes Zentrum Nordrhein-Westfalen, Oeyenhausen
  - Universitat Regensburg, Regensburg
  - Marienkrankenhaus Soest, Soest
  - Robert-Bosch-Krankenhaus, Stuttgart
- Italy (15):
  - Ospedale Civile S. Giuseppe, Albano Laziale
  - Azienda Ospedaliera S. Michele, Cagliari
  - Ospedale Civile, Capri city
  - Azienda USL n. 6 Ospedale Civile, Cecina
  - Poliambulatorio Valdichiana Ospedale di Cortona, Cortona
  - Centro Cardiologico Monzino, Milan
  - Ospedale Nigaurda Ca Granda, Milan
  - Fondazione Salvatore Maugeri, Montescano
  - Presidio Ospedaliero Villa Sofia, Palmero
  - Ospedali Riunti, Parma
  - IRCCS Policlinico S. Matteo, Pavia
  - IRCCS- Fondazione Salvatore Maugeri, Pavia
  - Ospedale S. Maria delle Grazie, Pozzuoli
  - Ospedale S. Bartolomeo, Sarzana
  - Ospedali Civile SS Annunziata, Sassari
- Netherlands (14):
  - Jeroen Bosch Ziekenhus (location Groot Ziekengasthius=GZG), 's-Hertogenbosch
  - Sint Lucas Andreas Ziekenhuis (loc. Lucas), Amsterdam
  - Gelre Ziekenhuis (location Juliana), Apeldoorn
  - Ziekenhuis Gooi Noord, Blaricum
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
  - Oosterschelde Ziekenhuizen, Goes
  - Martini Ziekenhuis (Loc. Martini Paviljoen), Groningen
  - Spaarne Ziekenhuis, Heemstede
  - Ziekenhuis Hilversum, Hilversum
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Medisch Centrum Haaglanden (location Westeinde), The Hague
  - Isala Klinieken (Loc. Sophia), Zwolle
- Norway (6):
  - Hjerte med. Avd. Haukeland Universitets Sykehus, Bergen
  - Nordlandsykehuset, Bodø
  - Hjertemed.avd. Akershus Universitetssykenhus, Nordbyhagen
  - Diakonhjemmets sykehus Oslo, Oslo
  - Med. Avd. Sykenhuset Telemark, Skien
  - Stavanger Helseforskning, Stavanger
- Poland (14):
  - Oddzial Kardiologii, Bydgoszcz
  - Oddzial Kardiologii, Krakow
  - Oddzial Kardiologii, Lodz
  - Oddzial Kardiologiczny, Opole
  - Oddzial Kardiologii, Ostrowiec Świętokrzyski
  - Oddzial Chorob Wewnetrznych, Oława
  - Oddzial Kardiologiczny, Piotrkow Trybunalski
  - Oddzial Kardiologiczny, Płock
  - Oddzial Kardiologii, Sieradz
  - Oddzial Kardiologii, Torun
  - Katedra i Oddzial Kliniczny Kardiologii Slaskiej Akademii, Tychy
  - I Klinika Choroby Wiencowej, Warsaw
  - Katedra i Klinika Chorab Wewnetrznych i Kardiologii, Warsaw
  - Oddzial Kardiologii, Włocławek
- Romania (11):
  - Spitalul Judetean Brasov, Sectia de Cardiologie, Brasov
  - Institutul de Boli Cardiovasculare, Bucharest
  - Spitalul Caritas, Clinica Medicala, Bucharest
  - Spitalul de Urgenta Floreasca, Clinica de Cardiologie, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Universitar de Urgenta, Bucharest
  - Institutul Inimii, Prof.N. Stancioiu, Cluj-Napoca
  - Centrul de Cardiologie Craiova, Craiova
  - Spitalul Clinic Universitar ,,Sf. Spiridon", Iași
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Institutul de Boli Cardiovasculare Timisoara, Timișoara
- Russia (24):
  - Botkins Moscow City Hospital, Moscow
  - Burdenko Main Military Clinical Hospital, Moscow
  - Cardiology Research Center, Moscow
  - Central Clinical Hospital Presidential, Moscow
  - City Clinical Hospital 2, Moscow
  - Institute of Physico-Chemical Medicine, Moscow
  - Medical Center of General Management, Moscow
  - Moscow Medical Academy, Moscow
  - Moscow Regional Research Clinical Institute n.a. Vishnevsky, Moscow
  - Moscow State University of Medicine and Dentistry - City Hospital #11, Moscow
  - Moscow State University of Medicine and Dentistry - City Hospital #40, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - Russian State Medical University, Moscow
  - Veterans Hospital #3, Moscow
  - Cardiology Research Institute of the Ministry of Health of the Russian Federation, Saint Petersburg
  - City Alexandrovsky Hospital, ICU Department, Saint Petersburg
  - City Hospital #31, Saint Petersburg
  - City Hospital 8, Saint Petersburg
  - Military Medical Academy, Saint Petersburg
  - St. Elisabeth City Hospital, Saint Petersburg
  - St. Petersburg Clinical Hospital of Russian Academy of Sciences, Saint Petersburg
  - St. Petersburg Dzanelidze State Scientific Research Institute for Emergency Medical Care, Saint Petersburg
  - St. Petersburg Medical Postgraduate Academy, Saint Petersburg
  - St. Petersburg State University, Saint Petersburg
- Spain (8):
  - Hospital de Torrecardenas, Almería
  - Hospital Clinic y Provincial, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Reina Sofia, in Cordoba, Córdoba
  - Hospital Doce de Octubre, Madrid
  - Hospital Severo Ochoa, Madrid
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital General Universitario de Valencia, Valencia
- Sweden (10):
  - Avd. for intermedicin, Gothenburg
  - Medicinkliniken, Gothenburg
  - Kardiologkliniken, Linköping
  - Kardiologkliniken, Malmo
  - Forskiningsenheten,, Mölndal
  - Enheten for internmedicin, Karolinska Institutet, Stockholm
  - Hjartkliniken, M84, Stockholm
  - Kardiologkliniken, Stockholm
  - Hjartcentrum,, Umeå
  - Cardiologkliniken, Avd 50F, Uppsala
- Cardiocentro Ticino, Lugano, Switzerland
- United Kingdom (5):
  - Bradford Royal Infirmary, Bradford
  - Castle Hill Hospital, Cottingham
  - Leeds General Infirmary, Leeds
  - Northern Manchester General Hospital, Manchester
  - Scunthorpe General Hospital, Scunthorpe

REFERENCES:
- [Derived] Oka T, Tighiouart H, McCallum W, Tuttle M, Isaka Y, Konstam MA, Udelson JE, Sarnak MJ. Thresholds of Kidney Function Decline and Congestion Status and Their Relation with Outcomes among Discharged Heart Failure Patients. Clin J Am Soc Nephrol. 2025 Jul 11;20(9):1215-1225. doi: 10.2215/CJN.0000000768. PMID 40643971
- [Derived] Hejjaji V, Tang Y, Coles T, Jones PG, Reeve BB, Mentz RJ, Spatz ES, Dunlay SM, Caldwell B, Saha A, Tarver ME, Tran A, Patel KK, Henke D, Pina IL, Spertus JA. Psychometric Evaluation of the Kansas City Cardiomyopathy Questionnaire in Men and Women With Heart Failure. Circ Heart Fail. 2021 Sep;14(9):e008284. doi: 10.1161/CIRCHEARTFAILURE.120.008284. Epub 2021 Sep 1. PMID 34465123
- [Derived] Ter Maaten JM, Valente MA, Damman K, Cleland JG, Givertz MM, Metra M, O'Connor CM, Teerlink JR, Ponikowski P, Bloomfield DM, Cotter G, Davison B, Subacius H, van Veldhuisen DJ, van der Meer P, Hillege HL, Gheorghiade M, Voors AA. Combining Diuretic Response and Hemoconcentration to Predict Rehospitalization After Admission for Acute Heart Failure. Circ Heart Fail. 2016 Jun;9(6):e002845. doi: 10.1161/CIRCHEARTFAILURE.115.002845. PMID 27266853
- [Derived] Ambrosy AP, Khan H, Udelson JE, Mentz RJ, Chioncel O, Greene SJ, Vaduganathan M, Subacuis HP, Konstam MA, Swedberg K, Zannad F, Maggioni AP, Gheorghiade M, Butler J. Changes in Dyspnea Status During Hospitalization and Postdischarge Health-Related Quality of Life in Patients Hospitalized for Heart Failure: Findings From the EVEREST Trial. Circ Heart Fail. 2016 May;9(5):e002458. doi: 10.1161/CIRCHEARTFAILURE.115.002458. PMID 27140204
- [Derived] Mentz RJ, Greene SJ, Ambrosy AP, Vaduganathan M, Subacius HP, Swedberg K, Maggioni AP, Nodari S, Ponikowski P, Anker SD, Butler J, Gheorghiade M. Clinical profile and prognostic value of anemia at the time of admission and discharge among patients hospitalized for heart failure with reduced ejection fraction: findings from the EVEREST trial. Circ Heart Fail. 2014 May;7(3):401-8. doi: 10.1161/CIRCHEARTFAILURE.113.000840. Epub 2014 Apr 15. PMID 24737459
- [Derived] Hauptman PJ, Burnett J, Gheorghiade M, Grinfeld L, Konstam MA, Kostic D, Krasa HB, Maggioni A, Ouyang J, Swedberg K, Zannad F, Zimmer C, Udelson JE; Everest Investigators. Clinical course of patients with hyponatremia and decompensated systolic heart failure and the effect of vasopressin receptor antagonism with tolvaptan. J Card Fail. 2013 Jun;19(6):390-7. doi: 10.1016/j.cardfail.2013.04.001. Epub 2013 May 14. PMID 23743487
- [Derived] Ambrosy AP, Vaduganathan M, Mentz RJ, Greene SJ, Subacius H, Konstam MA, Maggioni AP, Swedberg K, Gheorghiade M. Clinical profile and prognostic value of low systolic blood pressure in patients hospitalized for heart failure with reduced ejection fraction: insights from the Efficacy of Vasopressin Antagonism in Heart Failure: Outcome Study with Tolvaptan (EVEREST) trial. Am Heart J. 2013 Feb;165(2):216-25. doi: 10.1016/j.ahj.2012.11.004. Epub 2012 Dec 29. PMID 23351825
- [Derived] Allen LA, Gheorghiade M, Reid KJ, Dunlay SM, Chan PS, Hauptman PJ, Zannad F, Konstam MA, Spertus JA. Identifying patients hospitalized with heart failure at risk for unfavorable future quality of life. Circ Cardiovasc Qual Outcomes. 2011 Jul;4(4):389-98. doi: 10.1161/CIRCOUTCOMES.110.958009. Epub 2011 Jun 21. PMID 21693723
- [Derived] O'Connor CM, Miller AB, Blair JE, Konstam MA, Wedge P, Bahit MC, Carson P, Haass M, Hauptman PJ, Metra M, Oren RM, Patten R, Pina I, Roth S, Sackner-Bernstein JD, Traver B, Cook T, Gheorghiade M; Efficacy of Vasopressin Antagonism in heart Failure Outcome Study with Tolvaptan (EVEREST) investigators. Causes of death and rehospitalization in patients hospitalized with worsening heart failure and reduced left ventricular ejection fraction: results from Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study with Tolvaptan (EVEREST) program. Am Heart J. 2010 May;159(5):841-849.e1. doi: 10.1016/j.ahj.2010.02.023. PMID 20435194
- [Derived] Blair JE, Zannad F, Konstam MA, Cook T, Traver B, Burnett JC Jr, Grinfeld L, Krasa H, Maggioni AP, Orlandi C, Swedberg K, Udelson JE, Zimmer C, Gheorghiade M; EVEREST Investigators. Continental differences in clinical characteristics, management, and outcomes in patients hospitalized with worsening heart failure results from the EVEREST (Efficacy of Vasopressin Antagonism in Heart Failure: Outcome Study with Tolvaptan) program. J Am Coll Cardiol. 2008 Nov 11;52(20):1640-8. doi: 10.1016/j.jacc.2008.07.056. PMID 18992654
- [Derived] Gheorghiade M, Konstam MA, Burnett JC Jr, Grinfeld L, Maggioni AP, Swedberg K, Udelson JE, Zannad F, Cook T, Ouyang J, Zimmer C, Orlandi C; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study With Tolvaptan (EVEREST) Investigators. Short-term clinical effects of tolvaptan, an oral vasopressin antagonist, in patients hospitalized for heart failure: the EVEREST Clinical Status Trials. JAMA. 2007 Mar 28;297(12):1332-43. doi: 10.1001/jama.297.12.1332. Epub 2007 Mar 25. PMID 17384438
- [Derived] Konstam MA, Gheorghiade M, Burnett JC Jr, Grinfeld L, Maggioni AP, Swedberg K, Udelson JE, Zannad F, Cook T, Ouyang J, Zimmer C, Orlandi C; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study With Tolvaptan (EVEREST) Investigators. Effects of oral tolvaptan in patients hospitalized for worsening heart failure: the EVEREST Outcome Trial. JAMA. 2007 Mar 28;297(12):1319-31. doi: 10.1001/jama.297.12.1319. Epub 2007 Mar 25. PMID 17384437